CLINICAL TRIAL: NCT02153970
Title: The Calibration and Validation of the PROMIS and Neuro-QOL Questionnaires in Cerebral Palsy and Congenital Muscular Dystrophy
Brief Title: Calibration and Validation of the PROMIS and Neuro-QOL Questionnaires in Cerebral Palsy and Congenital Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140118; 14-NR-0118
Record Dates: First submitted 2014-05-31; First posted 2014-06-03 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06-12

CONDITIONS: Cerebral Palsy; Neuromuscular Disease
Keywords: Clinical Outcomes Measures; Proxy Reported Outcome; Pediatric; Neuromuscular Disease; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Neuromuscular diseases (NMDs) do not have cures. But future treatments will try to improve the health-related quality of life (HRQoL) in people with NMD. Computer questionnaires can help test HRQoL in people with NMD. They could help clinicians and researchers know how people with NMD and their caregivers are doing. They could also help show if treatments are making a difference.

Researchers want to make sure two of these questionnaires PROMIS (Patient Reported Outcomes Measurement Information System) and Neuro-QOL (Quality of Life in Neurological Disorders) work the same way every time. They also want to make sure the questionnaires test the same things every time.

Objective:

- To make sure the PROMIS and Neuro-QOL questionnaires are valid.

Eligibility:

- Children age 8 17 who have NMD. Also, caregivers of children age 5 17 who have NMD.

Design:

* Participants will complete the PROMIS and Neuro-QOL questionnaires on a computer. The caregiver and child versions are not the same.
* Participants will complete the questionnaires at the beginning of the study. It will take about 15 20 minutes. They will complete the questionnaires again after 2 4 weeks. They may receive phone or email reminders.
* Participants will complete the questionnaires at the NIH outpatient clinic and/or on their own device. At NIH, they will use a computer or tablet.

DETAILED DESCRIPTION:
Health-related quality of life (HRQoL) is defined as an individual s perception of his or her well-being and satisfaction with their current circumstances. As is oftentimes the case, in childhood-onset neuromuscular disease (NMD) and cerebral palsy (CP), no definitive cures currently exist. As a result, the primary goal of treatment for these patient populations is to improve quality of life or, more specifically, HRQoL. The medical community s interest in patient-based outcomes such as HRQoL has increased in the last two decades as it allows a multidimensional consideration of a patient s health. This focus has been the impetus for the development of computerized adaptive testing (CAT) instruments such as Quality of Life in Neurological Disorders (Neuro-QOL) and Patient Reported Outcomes Measurement Information System (PROMIS) to provide a means of assessing quality of life in patient populations with chronic diseases, such as neuromuscular disease and cerebral palsy.

The objective of this study is thus to validate the PROMIS and Neuro-QOL scales pediatric domains of self-assessment for individuals with CP and NMD and the PROMIS proxy domains for proxy-assessment of the same populations. The questionnaires will be administered to a combined total of 650 individuals from two sites in order to also calibrate the items and convert the questionnaires into CAT format.

The study population is patients with CP or NMD, ages 8-17 years, caregivers of patients with CP or NMD, whose children are ages 5-17 years. Caregivers are defined in this study as parents or legal guardians of children.

<TAB>

The design is a prospective study in which patients and caregivers will complete online versions of the PROMIS and Neuro-QOL questionnaires at one of two different sites.

<TAB>

The outcome measures are the responses to the questionnaires.

<TAB>

The validation of self-report and proxy-report questionnaires for use in the pediatric population with childhood-onset disease, specifically CP and NMD, will serve as an adjunct to the clinical exam and provide a way for clinicians and researchers to track the effectiveness of regular care and surgical interventions in these populations. The ultimate goal is to produce reliable, validated assessments of HRQoL in these populations via the CAT testing format with the potential to use these tools to inform both clinical decision-making and further research efforts for patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Children 8-17 years old who have been diagnosed with a neuromuscular disorder.
* Caregivers of children 5-17 years old diagnosed with a neuromuscular disorder.
* Caregivers have primary responsibility for the care of the child.
* All participants must be able to read English fluently.
* Caregivers are able to give consent for themselves and/or their child.

EXCLUSION CRITERIA:

-Caregivers may not be eligible for this research study if they become distressed when talking about their child s illness.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-05-31; Primary Completion 2018-04-04 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Responses to NeuroQol and PROMIS questionnaires | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Katherine G Meilleur, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gershon RC, Lai JS, Bode R, Choi S, Moy C, Bleck T, Miller D, Peterman A, Cella D. Neuro-QOL: quality of life item banks for adults with neurological disorders: item development and calibrations based upon clinical and general population testing. Qual Life Res. 2012 Apr;21(3):475-86. doi: 10.1007/s11136-011-9958-8. Epub 2011 Aug 27. PMID 21874314
- [Background] Cella D, Riley W, Stone A, Rothrock N, Reeve B, Yount S, Amtmann D, Bode R, Buysse D, Choi S, Cook K, Devellis R, DeWalt D, Fries JF, Gershon R, Hahn EA, Lai JS, Pilkonis P, Revicki D, Rose M, Weinfurt K, Hays R; PROMIS Cooperative Group. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. J Clin Epidemiol. 2010 Nov;63(11):1179-94. doi: 10.1016/j.jclinepi.2010.04.011. Epub 2010 Aug 4. PMID 20685078
- [Background] Cella D, Nowinski C, Peterman A, Victorson D, Miller D, Lai JS, Moy C. The neurology quality-of-life measurement initiative. Arch Phys Med Rehabil. 2011 Oct;92(10 Suppl):S28-36. doi: 10.1016/j.apmr.2011.01.025. PMID 21958920